CLINICAL TRIAL: NCT01729182
Title: Nexium Capsules Specific Clinical Experience Investigation for Long-term Use Concerning Prevention of Recurrence of Gastric Ulcer or Duodenal Ulcer With LDA
Brief Title: Nexium Capsules LDA Specific Clinical Experience Investigation
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D961PC00002
Record Dates: First submitted 2012-11-14; First posted 2012-11-20 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Gastric Ulcer; Duodenal Ulcer
Keywords: Low dose Aspirin(LDA); Gastric ulcer or duodenal ulcer; Nexium
MeSH Terms: conditions — Stomach Ulcer; Duodenal Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Nexium

SUMMARY:
The purpose of this investigation is to collect following data in patients given Nexium capsule (Nexium) for long term in usual-post-marketing therapy to prevention of recurrence of gastric ulcer or duodenal ulcer with Low dose Aspirin (LDA).

DETAILED DESCRIPTION:
Nexium capsules Specific Clinical Experience Investigation for long-term use concerning prevention of recurrence of gastric ulcer or duodenal ulcer with Low dose Aspirin (LDA).

ELIGIBILITY:
Exclusion Criteria:

* Patients having gastric ulcer/duodenal ulcer when Nexium is started (Active phase (A1, A2) or healing phase (H1, H2) of Sakita-Miwa classification on endoscopy).
* Patients who had been given Nexium for suppression of recurrence of gastric ulcer/duodenal ulcer.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients who are continuously given Low dose Aspirin (LDA) to suppress thrombus/embolism and who will be given Nexium for the first time to suppress recurrence of gastric ulcer and duodenal ulcer.
  (Patients who have previous experience of Nexium given in the treatment for gastric ulcer or duodenal ulcer can be registered to this S-CEI.)
Sampling Method: Non-Probability Sample
Enrollment: 2363 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2017-03-09 (Actual); Study Completion 2017-03-09 (Actual)

PRIMARY OUTCOMES:
Adverse events incidence | Up to 2 years
  Number of Adverse Drug Reactions

SECONDARY OUTCOMES:
Non-recurrence rate of peptic ulcer | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Shigeru Yoshida, MD, Study Director — AstraZeneca
Locations (47):
- Japan (47):
  - Research Site, Aichi
  - Research Site, Akita
  - Research Site, Aomori
  - Research Site, Chiba
  - Research Site, Ehime
  - Research Site, Fukui
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Gifu
  - Research Site, Gunma
  - Research Site, Hiroshima
  - Research Site, Hokkaido
  - Research Site, Hyōgo
  - Research Site, Ibaraki
  - Research Site, Ishikawa
  - Research Site, Kagawa
  - Research Site, Kagoshima
  - Research Site, Kanagawa
  - Research Site, Kochi
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Mie
  - Research Site, Miyagi
  - Research Site, Miyazaki
  - Research Site, Nagano
  - Research Site, Nagasaki
  - Research Site, Nara
  - Research Site, Niigata
  - Research Site, Numakunai
  - Research Site, Okayama
  - Research Site, Okinawa
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Saga
  - Research Site, Saitama
  - Research Site, Shiga
  - Research Site, Shimane
  - Research Site, Shizuoka
  - Research Site, Tochigi
  - Research Site, Tokushima
  - Research Site, Tokyo
  - Research Site, Tottori
  - Research Site, Toyama
  - Research Site, Wakayama
  - Research Site, Yamagata
  - Research Site, Yamaguchi
  - Research Site, Yamanashi

REFERENCES:
- See also: AZ_Synopsis_D961PC00002 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=709&filename=AZ%20Synopsis%20_D961PC00002.pdf
- See also: K. Sakamoto, M. Nii, T. Tokimoto and Y. Takumi Efficacy and Safety of Esomeprazole (Nexium) for the Prevention of Recurrent Gastric or Duodenal Ulcers in Patients on Continuous LDA; PMS of Long-term Use Jpn Pharmacol Ther, 47(6), 893 - 910, 2019 — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D961PC00002&attachmentIdentifier=3369ebc0-0d02-4d61-998f-b9321c317c64&fileName=NEX_SCEI_LDA_Protocol(E)_Ver3_redacted.pdf&versionIdentifier=